CLINICAL TRIAL: NCT03289845
Title: Clinical Survey of Oticon Medical Ponto BHX Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C55
Record Dates: First submitted 2017-08-31; First posted 2017-09-21 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Hearing Impaired (Partially); Hearing Impairment, Conductive; Deafness Unilateral
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BHX implant (Other): All patients implanted with BHX implant
  Interventions: Device: BHX implant (Bone anchored hearing system)

INTERVENTIONS:
Device: BHX implant (Bone anchored hearing system) — Bone anchored hearing system for hearing rehabilitation

SUMMARY:
Investigation of stability of the BHX implant in adult patients indicated and counselled for a bone anchored hearing aid system. Patients are followed according to clinical practice for a total of 12 months in the study. Stability of the implant is evaluated by implant stability quotient.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for treatment with a bone anchored hearing aid
* 18 years or older

Exclusion Criteria:

* Inability to participate in follow-up
* Diseases or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Implant stability quotient (ISQ) at surgery | At surgery
  Initial implant stability measured directly after surgery

SECONDARY OUTCOMES:
Surgical torque setting measured in Ncm | At surgery
  The surgical torque setting used to install the implant
Possibility to fit the sound processor, yes/no | 5-12 days post surgery
  Fitting of the sound processor at 5-12 days post-surgery
Implant stability quotient (ISQ) after 12 months of follow up | 12 months post surgery
  Long term stability development
Implant survivability measured as percentage successful implants after 12 months | 12 months post surgery
  Implant survivability

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Dept. of Otolaryngology - Head & Neck Surgery and Audiology, Gentofte/Rigshospitalet,, Hellerup, Copenhagen
  - Department of Oto-Rhino-Laryngology & Audiology Aalborg University Hospital, Aalborg

IPD SHARING:
Plan to Share IPD: No